CLINICAL TRIAL: NCT00082862
Title: A Phase II Clinical Trial of a Timing/Schedule Optimized Combined-Modality Regimen: Cisplatin + Metronomic Low-Dose Interferon-α (IFN-α) Followed by Gemcitabine HCl (GEMZAR) in Combination With Mild, Fever-Range Whole-Body Hyperthermia (FR-WBH) in Patients With Advanced, Inoperable Pancreatic Cancer
Brief Title: Cisplatin, Metronomic Low-Dose Interferon Alfa, Gemcitabine, and Fever-Range Whole-Body Hyperthermia in Treating Patients With Inoperable or Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Joan M.C. Bull, University of Texas Health Science Center at Houston
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000360863; UTHSC-MS-02117
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2008-12

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Interferon-alpha; Cisplatin; Gemcitabine; Diathermy

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving low-dose interferon alfa on a metronomic (regularly timed) schedule may stop the growth of cancer by stopping blood flow to the tumor. Fever-range (above 101° F) whole-body hyperthermia kills tumor cells by heating them to several degrees above normal body temperature. Combining cisplatin, gemcitabine, and low-dose interferon alfa with fever-range whole-body hyperthermia may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin, gemcitabine, and metronomic low-dose interferon alfa together with fever-range whole-body hyperthermia works in treating patients with inoperable or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine tumor response in patients with inoperable or metastatic pancreatic cancer treated with cisplatin, metronomic low-dose interferon alfa, gemcitabine, and fever-range whole-body hyperthermia.
* Determine the toxicity of this regimen in these patients.
* Determine the survival of patients treated with this regimen.
* Determine changes in quality of life in patients treated with this regimen.

Secondary

* Determine whether inoperable tumors convert to operable in patients treated with this regimen.
* Determine changes in cellular and cytokine immune function in patients treated with this regimen.

OUTLINE: Patients are stratified according to disease stage (metastatic vs inoperable).

Patients receive cisplatin IV over 4-6 hours on day 1, interferon alfa subcutaneously once daily on days 1-28, and gemcitabine IV over 1 hour on days 3 and 10. Patients undergo fever-range whole-body hyperthermia (40°C over 6 hours) on day 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then before each treatment course.

PROJECTED ACCRUAL: A total of 18-48 patients (9-24 per stratum) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic carcinoma

  * Inoperable or metastatic disease
* Measurable lesion by physical examination, CT scan, or MRI

  * Carcinomatous hepatomegaly is considered measurable if a palpable liver edge clearly extends > 15 cm below the costal margin or xiphoid process
* No known brain metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin > 10.0 g/dL
* Platelet count ≥ 90,000/mm^3
* Bone marrow cellularity normal on bone marrow biopsy
* No serious coagulopathy disorder

Hepatic

* Bilirubin ≤ 2.5 mg/dL
* SGPT and SGOT ≤ 2 times upper limit of normal
* PT < 14 seconds
* PTT < 35 seconds
* INR < 1.5

Renal

* Creatinine ≤ 1.8 mg/dL
* Creatinine clearance ≥ 45 mL/min
* Blood urea nitrogen ≤ 25 mg/dL

Cardiovascular

* Adequate cardiovascular function as documented by the following:

  * History and physical examination
  * Stress exercise test (MUGA or echocardiogram) with resting blood pressure, heart rate, and LVEF that increase appropriately with exercise
  * LVEF ≥ 45%
* No myocardial infarction within the past 6 months
* No symptomatic coronary artery disease
* No angina
* No unstable blood pressure
* No congestive heart failure
* No significant arrhythmia
* No conduction disturbance
* No thromboembolic disease
* No uncontrolled hypertension

Pulmonary

* Complete pulmonary function studies with the following arterial blood gas values:

  * FEV_1 ≥ 70% of predicted
  * Arterial PO_2 ≥ 60 mm Hg on room air
  * PCO_2 appropriate
  * pH appropriate
* No massive (≥ 30%) lung disease
* DLCO > 50% of predicted

Other

* No prior or concurrent seizures or other CNS disorders
* No prior malignant hyperthermia after general anesthesia
* No insulin-dependent diabetes mellitus
* No significant emotional instability
* No other medical problem that would preclude treatment with whole-body hyperthermia
* HIV negative
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed

Chemotherapy

* No prior cisplatin or gemcitabine

Endocrine therapy

* No concurrent adrenal corticosteroids

Radiotherapy

* More than 3 weeks since prior radiotherapy

Surgery

* More than 6 days since prior major thoracic or abdominal surgery
* Prior surgical resection of tumor with subsequent recurrence allowed

Other

* No concurrent cardiac glycosides
* No concurrent anti-angina or arrhythmia drugs
* No concurrent thrombolytic agents
* No concurrent anticoagulants
* No concurrent aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2002-07; Primary Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Tumor response
Toxicity
Survival
Changes in quality of life

SECONDARY OUTCOMES:
Conversion of inoperable tumors to operable
Changes in cellular and cytokine immune function

CONTACTS AND LOCATIONS:
Overall Officials: Joan M.C. Bull, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Bull JM, Scott GL, Strebel FR, Nagle VL, Oliver D, Redwine M, Rowe RW, Ahn CW, Koch SM. Fever-range whole-body thermal therapy combined with cisplatin, gemcitabine, and daily interferon-alpha: a description of a phase I-II protocol. Int J Hyperthermia. 2008 Dec;24(8):649-62. doi: 10.1080/02656730802104740. PMID 18608594